CLINICAL TRIAL: NCT01164306
Title: The Impact of a Tobacco Control Intervention in African-American Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Martha Tingen, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA118066 (NIH); R01CA118066 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-07-16 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Tobacco Prevention; Environmental Tobacco Smoke Exposure; Tobacco Cessation
Keywords: LifeSkills Training; Tobacco prevention; Tobacco cessation; Healthy lifestyles; Tobacco control
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Nicotine Replacement Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LifeSkills training (Experimental)
  Interventions: Behavioral: LifeSkills Training; Behavioral: NRT and Motivational Interviewing (MI)
- Healthy Lifestyle Behaviors (Active Comparator)
  Interventions: Behavioral: Healthy Lifestyle Behavior Choices

INTERVENTIONS:
Behavioral: LifeSkills Training — LifeSkills Training (Botvin's) is an evidenced based substance abuse prevention program for elementary school students to learn skills to resist tobacco, alcohol, drug abuse, and violence.
  Parent LifeSkills will also be utilized. Parents are provided a parent manual and DVD to use at home with their child to reinforce what they are taught in school-based LifeSkills sessions.
  Other Names: LifeSkills Training (Botvin's)
  Arms: LifeSkills training
Behavioral: Healthy Lifestyle Behavior Choices — The healthy lifestyle behavior choices curriculum augments the state health curriculum in the assigned study schools.
  Parents will also be given health related information by mail to parallel the information students receive in school health classes.
  Other Names: Healthy lifestyle behaviors
  Arms: Healthy Lifestyle Behaviors
Behavioral: NRT and Motivational Interviewing (MI) — For parent/guardian smokers who want to quit, NRT is offered in conjunction with MI.
  Other Names: NRT is Nicotine Replacement Therapy; MI is Motivational Interviewing
  Arms: LifeSkills training

SUMMARY:
The purpose of this randomized control trial is to evaluate the effects of a multi-component intervention aimed at:

1. preventing tobacco initiation in youth
2. promoting anti-tobacco socialization in the home
3. decreasing environmental tobacco smoke exposure in children
4. promoting successful cessation in parent/guardian smokers.

Control arm participants receive general health education. This family-based approach is implemented with school systems as the primary point of entry.

DETAILED DESCRIPTION:
All research participants (children and parents/guardians) will be recruited from 14 schools (7 control and 7 intervention; 7 urban and 7 rural) in a Southeastern U.S.

Self-report measures are at: baseline, end of year one, year 2, end of year two, and years three and four. Biological measures of salivary cotinine are at Baseline, end of treatment (year 2) and end of study (year 4).

ELIGIBILITY:
Inclusion Criteria:

* child being of African-American ethnicity
* in a 4th grade classroom of randomized schools
* parent or guardian that 4th grade child resides with at least 50% of the time
* have access to a telephone or mobile phone

Exclusion Criteria:

* not being a child of African-American ethnicity
* not being a parent or guardian that an eligible child lives with at least 50% of the time
* not having access to a telephone or cell phone

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2007-09; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Primary prevention of tobacco use in youth | Baseline
  Self-report and salivary cotinine is assessed to measure this outcome
Primary prevention of tobacco use in youth | Year 2
  Self-report and salivary cotinine is assessed to measure this outcome.
Primary prevention of tobacco use in youth | Year 4
  Self-report and salivary cotinine is assessed to measure this outcome.

SECONDARY OUTCOMES:
Smoking cessation in parents/guardians | 3 months
Smoking cessation in parents/guardians | 6 months
Smoking cessation in parents/guardians | Year 1
Smoking cessation in parents/guardians | Year 2
Smoking cessation in parents/guardians | Year 4

CONTACTS AND LOCATIONS:
Overall Officials: Martha S Tingen, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Caldwell AL, Tingen MS, Nguyen JT, Andrews JO, Heath J, Waller JL, Treiber FA. Parental Smoking Cessation: Impacting Children's Tobacco Smoke Exposure in the Home. Pediatrics. 2018 Jan;141(Suppl 1):S96-S106. doi: 10.1542/peds.2017-1026M. PMID 29292310